CLINICAL TRIAL: NCT04379323
Title: Validation of the YuWell YE900 Medical Electronic Blood Pressure Monitor in Adults and Children According to the AAMI/ESH/ISO 81060-2:2018 Standard
Brief Title: Clinical Trial of YuWell YE900 Electronic Sphygmomanometer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Collaborators: Jiangsu Yuyue medical equipment & supply Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, zhang Hui Jie, Director of Clinical trial center, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: YUWELL-YLQX202001
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Blood Pressure
Keywords: AAMI/ESH/ISO 81060-2: 2018 standard; blood pressure measurement; blood pressure monitor; validation study; YuWell YE900
MeSH Terms: interventions — Blood Pressure Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YuWell YE900 and mercury sphygmomanometer (Experimental): Blood Pressure Measurement with the YuWell YE900 Electronic Sphygmomanometer (YuWell YE900) and with Desk Mercury Sphygmomanometer.
  Interventions: Diagnostic Test: YuWell YE900 Electronic Sphygmomanometer

INTERVENTIONS:
Diagnostic Test: YuWell YE900 Electronic Sphygmomanometer — Measurement blood pressure by YuWell YE900 Electronic Sphygmomanometer and Desk Mercury Sphygmomanometer.
  Other Names: Desk Mercury Sphygmomanometer; Blood Pressure Measurement

SUMMARY:
The purpose of this study is to evaluate the accuracy of the YuWell YE900 medical electronic blood pressure monitor for blood pressure measurements in adults and children according to the Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO) Universal Standard (ISO 81060-2:2018).

ELIGIBILITY:
Inclusion Criteria:

1. 3 Years and older (Child, Adult, Older Adult);
2. Subjects voluntarily participate in the clinical trial and sign the informed consent.

Exclusion Criteria:

1. Disturbance of consciousness;
2. Patients requiring hemodialysis;
3. Taking anticoagulant drugs due to cardiovascular and cerebrovascular diseases;
4. Pregnant and lactating women;
5. Patients with cardiac arrhythmias;
6. Other conditions that the investigator considers ineligible for clinical trial.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurement data | 30 minutes
  Systolic Pressure and Diastolic Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi Long, MD PHD, Study Director — The Second Hospital of Nanjing Medical University
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang HJ, Zhang J, Wang SL, Zhang J, Teng LN, Zhang SJ, Zhou DJ, Long MZ. Validation of the YuWell YE900 oscillometric blood pressure monitor for professional office use in adults and children according to the AAMI/ESH/ISO Universal Standard (ISO 81060-2:2018). Blood Press Monit. 2021 Oct 1;26(5):396-399. doi: 10.1097/MBP.0000000000000541. PMID 34480474